CLINICAL TRIAL: NCT05876715
Title: LINNOVATE: A Phase 1/2 Study of Safety/Efficacy Using LURBINECTEDIN, Combined With IPILIMUMAB, and NIVOLUMAB for Advanced Soft Tissue Sarcomas
Brief Title: LINNOVATE: Lurbinectedin, Ipilimumab and Nivolumab for Soft Tissue Sarcoma
Acronym: LINNOVATE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ERLINDA M GORDON (Other)
Responsible Party: Sponsor-Investigator, ERLINDA M GORDON, Director, Gene and Cell Therapy/Immunotherapy, Sarcoma Oncology Research Center, LLC
Organization: Sarcoma Oncology Research Center, LLC (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOC-2310
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Advanced Soft-tissue Sarcoma
MeSH Terms: interventions — PM 01183; Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is an open label, dose-seeking phase 1/2 study using escalating doses of LURBINECTEDIN administered intravenously with fixed doses of IPILIMUMAB and NIVOLUMAB administered intravenously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Phase 1/2 study using lurbinectedin, ipilimumab and nivolumab for advanced soft tissue sarcoma (Experimental): This is an open label, dose-seeking phase 1/2 study using escalating doses of LURBINECTEDIN administered intravenously with fixed doses of IPILIMUMAB and NIVOLUMAB administered intravenously.
  I. Dose Escalation Phase 1 of Study: The study will employ the standard "cohort of three" design (Storer, 1989).
  II.Phase 2 of Study: Following completion of dose escalation, an additional 28-34 previously untreated participants will receive LURBINECTEDIN at the MTD and fixed doses of IPILIMUMAB and NIVOLUMAB to assess overall safety and potential efficacy in a larger number of participants.
  Interventions: Drug: Lurbinectedin

INTERVENTIONS:
Drug: Lurbinectedin — This is an open label, dose-seeking phase 1/2 study using escalating doses of LURBINECTEDIN administered intravenously with fixed doses of IPILIMUMAB and NIVOLUMAB administered intravenously.
  Other Names: Ipilimumab; Nivolumab

SUMMARY:
This is an open label, dose-seeking phase 1/2 study using escalating doses of LURBINECTEDIN administered intravenously with fixed doses of IPILIMUMAB and NIVOLUMAB administered intravenously.

DETAILED DESCRIPTION:
This is an open label, dose-seeking phase 1/2 study using escalating doses of LURBINECTEDIN administered intravenously with fixed doses of IPILIMUMAB and NIVOLUMAB administered intravenously.

I. Dose Escalation Phase 1 of Study: The study will employ the standard "cohort of three" design (Storer, 1989). Three participants are treated at each of the 2 ascending dose levels. An additional 3 participants will be enrolled if a DLT is observed in one of the three initially-enrolled participants at each dose level. If no DLT occurs after the third participant in a dose level is on study for 6 weeks, enrollment will be opened for escalation to the next highest planned dose level. The DLT window is a total of 6 weeks. The MTD is defined as the highest safely tolerated dose of lurbinectedin, where not more than one participant experienced a DLT, with the next higher dose level having at least two participants who experienced DLT.

Participants in the dose escalation study may continue treatment at their designated dose levels until disease progression or unacceptable toxicity occurs or up to a maximum of one year of therapy (up to a maximum of 18 doses of LURBINECTEDIN, 26 doses of NIVOLUMAB, and 5 doses of IPILIMUMAB). No intra-participant dose escalation will take place.

Dose of IPILIMUMAB: 1 mg/kg IV over 30 min. q 12 weeks, beginning 2 weeks after the first dose of LURBINECTEDIN, until disease progression or unacceptable toxicity, up to a maximum of 5 doses

Dose of NIVOLUMAB: 3 mg/kg over 30 min. q 2 weeks, beginning 2 weeks after first dose of LURBINECTEDIN, until disease progression or unacceptable toxicity, up to a maximum of 26 doses

Dose of LURBINECTEDIN: Escalating doses of LURBINECTEDIN IV over 60 minutes q 3 weeks up to a maximum of 18 doses:

LURBINECTEDIN # Pts. Dose Level Dose,mg/m2 Max.Volume/24 hrs

Every 3 weeks 3-6 I 2.6 1000 ml Every 3 weeks 3-6 II 3.2 1000 ml

No dose-escalation will be performed until all the subjects have completed the DLT period of 6 weeks and evaluation of all clinical and laboratory data has been conducted. The phase 2 part of the study will not proceed until either the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been determined.

Participants who do not complete the DLT period for reasons other than study drug-related toxicity will be replaced in the same dose cohort. At the discretion of the principal investigator/sponsor, dose escalation may be stopped before an MTD is reached. In this case, the MAD may be chosen based on the standard dose of LURBINECTEDIN of 3.2 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the inclusion criteria in order to be eligible to participate in the study, as follows:

1. Male or Female ≥ 18 years of age
2. Pathologically confirmed diagnosis of locally advanced unresectable or metastatic soft tissue sarcoma
3. For the Phase 1 Part of Study, only previously treated participants will be enrolled. For the Phase 2 Part of Study, previously untreated participants will be enrolled.
4. Ability to understand the purposes and risks of the study and has signed and dated a written informed consent form approved by the principal investigator's IRB/Ethics Committee
5. Willingness to comply with all study procedures and availability for the duration of the study.
6. Measurable disease by RECIST v1.1
7. ECOG performance status ≤ 1
8. Life expectancy of at least 3 months

   1. Acceptable liver function: Bilirubin < 1.5 times upper limit of normal (ULN; except subjects with Gilbert Syndrome who must have a total bilirubin level < 3.0 ULN);
   2. AST (SGOT), ALT (SGPT) and alkaline phosphatase < 3 x ULN (< 5 x ULN if liver metastases)
   3. Acceptable renal function: Creatinine < 1.5 times ULN or > 60 mL/min (using the Cockcroft Gault formula)
9. Acceptable hematologic status (without hematologic support e.g. growth factors or transfusion within 21 days of first dose of study agents): ANC >= 1500 cells/μL; Platelet count >= 100,000/μL; Hemoglobin >= 9.0 g/dL; Normal PT, PTT, INR
10. All women of childbearing potential must have a negative pregnancy test and all subjects must agree to use highly effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 5 months for women and 7 months for men after the last dose.

Exclusion Criteria:

All individuals meeting any of the exclusion criteria at baseline will be excluded from study participation, as follows:

1. Subjects with untreated CNS metastases. Subjects are eligible if CNS metastases have been adequately treated and have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to treatment initiation. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of <10 mg daily prednisone (or equivalent) for at least 2 weeks prior to treatment initiation.
2. Subjects with carcinomatous meningitis
3. Anticancer treatment with radiation therapy, targeted therapy or other antitumor treatment within 2 weeks prior to study entry. Anticancer treatment with chemotherapy within 21 days prior to study entry.
4. Subjects who participated in an investigational drug or device study within 14 days prior to study entry
5. Females who are pregnant or breast-feeding
6. Unwillingness or inability to comply with the study protocol for any reason
7. Concurrent or prior immunotherapy with anti-CTLA4 or anti-PD-1 inhibitors
8. Non-oncology vaccine therapy used for prevention of infectious disease within 4 weeks of trial enrollment
9. Autoimmune disease including rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis and motor neuropathy considered to be of autoimmune origin (e.g. Guillain-Barre Syndrome)
10. Systemic immunosuppression, including HIV positive status with or without AIDS
11. Skin rash (psoriasis, eczema) affecting > 25% body surface area
12. Inflammatory bowel disease (Crohn's or ulcerative colitis)
13. Ongoing or uncontrolled diarrhea within 4 weeks of trial enrollment
14. Recent history of acute diverticulitis, intraabdominal abscess or gastrointestinal obstruction within 6 months of trial enrollment, which are known risk factors for bowel perforation
15. Participants with congestive heart failure or recent cardiac event
16. Evidence of severe or uncontrolled systemic disease or any other concurrent condition, including psychiatric, which in the principal investigator or sub-investigator's opinion makes it undesirable for the participant to participate in the trial or which would jeopardize compliance with the trial
17. Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
18. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
19. Current, active, or previous history of heavy alcohol abuse
20. Pituitary endocrinopathy
21. Adrenal insufficiency or excess

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 months
  The maximum tolerated dose (MTD) is defined as the highest safely tolerated dose of lurbinectedin, where not more than one participant experienced a dose limiting toxicity (DLT), with the next higher dose level having at least two participants who experienced DLT.

SECONDARY OUTCOMES:
Objective response rate | 24 months
  The number of patients achieving a complete response and partial response divided by the number of patients who completed at least one treatment cycle and had a follow up computerized tomography (CT) scan
Progression free survival at 6 months | 12 months
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Overall survival | 36 months
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive. I
Correlation of response with circulating tumor DNA | 36 months
  Correlation of response with circulating tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Erlinda M Gordon, MD, Principal Investigator — Sarcoma Oncology Research Center
Locations (1):
- Sarcoma Oncology Research Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
We have no plan to make individual participant data available to other researchers other than the Sarcoma Oncology Research Center team.

REFERENCES:
- [Background] Gordon EM, Chawla SP, Tellez WA, Younesi E, Thomas S, Chua-Alcala VS, Chomoyan H, Valencia C, Brigham DA, Moradkhani A, Quon D, Srikureja A, Wong SG, Tseng W, Federman N. SAINT: A Phase I/Expanded Phase II Study Using Safe Amounts of Ipilimumab, Nivolumab and Trabectedin as First-Line Treatment of Advanced Soft Tissue Sarcoma. Cancers (Basel). 2023 Jan 31;15(3):906. doi: 10.3390/cancers15030906. PMID 36765863
- [Background] Gordon EM, Sankhala KK, Chawla N, Chawla SP. Trabectedin for Soft Tissue Sarcoma: Current Status and Future Perspectives. Adv Ther. 2016 Jul;33(7):1055-71. doi: 10.1007/s12325-016-0344-3. Epub 2016 May 27. PMID 27234989
- [Background] Belgiovine C, Bello E, Liguori M, Craparotta I, Mannarino L, Paracchini L, Beltrame L, Marchini S, Galmarini CM, Mantovani A, Frapolli R, Allavena P, D'Incalci M. Lurbinectedin reduces tumour-associated macrophages and the inflammatory tumour microenvironment in preclinical models. Br J Cancer. 2017 Aug 22;117(5):628-638. doi: 10.1038/bjc.2017.205. Epub 2017 Jul 6. PMID 28683469
- [Background] Cespedes MV, Guillen MJ, Lopez-Casas PP, Sarno F, Gallardo A, Alamo P, Cuevas C, Hidalgo M, Galmarini CM, Allavena P, Aviles P, Mangues R. Lurbinectedin induces depletion of tumor-associated macrophages, an essential component of its in vivo synergism with gemcitabine, in pancreatic adenocarcinoma mouse models. Dis Model Mech. 2016 Dec 1;9(12):1461-1471. doi: 10.1242/dmm.026369. Epub 2016 Oct 20. PMID 27780828